CLINICAL TRIAL: NCT04206930
Title: Impact of Art Therapy on Alexithymia in People With Alcohol Use Disorder
Acronym: ALEXART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A02031-52
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Alexithymia; Alcohol Use Disorder
MeSH Terms: conditions — Affective Symptoms; Alcoholism | interventions — Art Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard support: information on alcoholic pathology, medico-psycho-social assessment, relapse prevention program
- Art-Therapy (Experimental): in addition to standard treatment, art therapy treatment program: 1 session of 2 hours per week in a closed group for 10 weeks
  Interventions: Other: Art Therapy

INTERVENTIONS:
Other: Art Therapy — 1 session of 2 hours per week in a closed group for 10 weeks
  Arms: Art-Therapy

SUMMARY:
Art therapy support combined with standard care for people with an alcohol use disorder coming to a day hospital for withdrawal could be beneficial compared to standard care alone because it would improve the alexithymia of these patients, helping them to better identify their feelings and / or emotions, and improve their self-confidence, their self-esteem self and their oral communication.

DETAILED DESCRIPTION:
Alexithymia is an inability to identify and describe one's emotions associated with outward thinking. Frequently found in people with an alcohol use disorder, a true mental handicap, alexithymia has been clearly identified as a relapse factor in addictive problems related to alcohol. The ALEXART study intends to study the evolution of alexithymia in people with an alcohol use disorder hosted in an Addictology Day Hospital unit through the use of an approach non-drug that is art therapy. Our hypothesis is that art therapy can help patients with alcohol use disorders to develop a better understanding of their own behaviors, to name their emotions and feelings, and to improve their communication with others and thereby be able to choose to change their behavior.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 or over
* Patient with an alcohol use disorder starting day hospital care in the psychiatry and addiction department of the Angers University Hospital
* Subjects who gave and signed informed consent to participate in the study with alexithymia (Toronto Test greater than or equal to 56)

Exclusion Criteria:

* Non-understanding of the French language
* Non-affiliation to a social security scheme
* Major cognitive impairment
* Motor problems preventing walking
* Protective patients
* Pregnant or lactating women
* Patients under protection of justice or deprived of liberty
* Patients under protective supervision or guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-01-07 (Estimated); Study Completion 2022-12-13 (Estimated)

PRIMARY OUTCOMES:
Echelle de Toronto (TAS) | 3 month after inclusion
  self-questionnaire which includes 20 items and allows to measure 3 factors:
  * Difficulty identifying feelings (TAS 1).
  * Difficulty expressing feelings (TAS 2).
  * Outward-oriented thinking (TAS 3).

CONTACTS AND LOCATIONS:
Overall Officials: BENEDICTE GOHIER, Study Director — CHU ANGERS SERVICE DE PSYCHIATRIE ADDICTOLOGIE
Locations (1):
- Centre Hospitalier Universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: No